CLINICAL TRIAL: NCT02360787
Title: The Effects of Including Almonds in an Energy-restricted Diet on Weight, Abdominal Fat Loss, Blood Pressure, and Cognitive Function
Brief Title: The Effects of Including Almonds in a Weight Loss Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Almond Board of California (Other)
Responsible Party: Principal Investigator, Richard Mattes, Distinguished Professor Nutrition Science, Purdue University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 055-030
Record Dates: First submitted 2014-11-20; First posted 2015-02-11 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Overweight; Obesity
Keywords: Almonds; Energy restriction; Obesity; Body weight; Body fat; Blood pressure; Cognitive function
MeSH Terms: conditions — Overweight; Obesity; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Energy restriction (Experimental): Energy restriction (-500 kcal/day) (N=40), where participants will receive dietary counseling to reduce energy intake to achieve 500 kcal/day deficits to support weight loss. Participants will also be asked to avoid all nuts during the intervention period.
  Interventions: Behavioral: Energy restriction
- Energy restriction with almonds (Experimental): Energy restriction (-500 kcal/day) with dry-roasted, lightly salted almonds supplying 15% of estimated energy requirement. Participants will receive dietary counseling to reduce energy intake to achieve 500 kcal/day deficits. Energy from almonds will be accounted for during dietary modeling so that a 500 kcal/day deficit is achieved.
  Interventions: Behavioral: Energy restriction; Behavioral: Almonds (15% kcal/day)

INTERVENTIONS:
Behavioral: Energy restriction
Behavioral: Almonds (15% kcal/day)
  Arms: Energy restriction with almonds

SUMMARY:
The purpose of this study is to determine whether inclusion of almonds in a weight loss regimen will augment the rate of weight loss, promote a greater fat mass/fat-free mass ratio of weight loss, improve blood pressure and ameliorate the post-lunch dip in cognitive function.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether inclusion of almonds in a weight loss regimen will augment the rate of weight loss, promote a greater fat mass/fat-free mass ratio of weight loss, improve blood pressure and ameliorate the post-lunch dip in cognitive function.

ELIGIBILITY:
Inclusion Criteria:

Adult participants

* Overweight or obese (BMI 25-40 kg/m2)
* Fasting blood glucose ≤6.9 mmol/L via capillary finger-stick blood samples
* No nut allergies
* Willing to comply to study protocol and to eat test meals

Exclusion Criteria:

Those not meeting inclusion criteria.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-10 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Anthropometric measurements | 12 weeks
  Changes in body weight, BMI, fat mass, waist circumference and abdominal height over 12 weeks
Blood pressure | 12 weeks
  Blood pressure measurements assessed at baseline, week-4, week-8 and week-12
Post-lunch cognitive function | 12 weeks
  Cognitive function assessments will be performed after a standard lunch at baseline and week 12

SECONDARY OUTCOMES:
Fasting blood biochemistries | 12 weeks
  Fasting glucose, insulin, lipids and vitamin E over 12 weeks
Dietary intake | 10 weeks
  Dietary intakes assessed at baseline, week-1, week-2, week-3, week-4, week-6, week-8 and week-10
Appetite ratings | 12 weeks
  Appetite ratings assessed at baseline, week-4, week-8 and week-12
Physical activity | 12 weeks
  Physical activity assessed at baseline, week-4, week-8 and week-12

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

REFERENCES:
- [Derived] Dhillon J, Ferreira CR, Sobreira TJP, Mattes RD. Multiple Reaction Monitoring Profiling to Assess Compliance with an Almond Consumption Intervention. Curr Dev Nutr. 2017 Sep 6;1(9):e001545. doi: 10.3945/cdn.117.001545. eCollection 2017 Sep. PMID 29955720
- [Derived] Dhillon J, Tan SY, Mattes RD. Almond Consumption during Energy Restriction Lowers Truncal Fat and Blood Pressure in Compliant Overweight or Obese Adults. J Nutr. 2016 Dec;146(12):2513-2519. doi: 10.3945/jn.116.238444. Epub 2016 Nov 2. PMID 27807041